CLINICAL TRIAL: NCT04520464
Title: Non-inferiority Clinical Trial Comparing the Self-test for Cervicovaginal Sample Versus Sample Collection by the Service Provider for the Identification of HPV-RA DNA and Triage With p16 & ki67 Dual Staining.
Brief Title: Clinical Trial Comparing the Self-test for Cervicovaginal Sample Versus Samples From Service Provider (Xyto-Ro)
Acronym: Xyto-Ro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Dr. Carlos E. Aranda Flores, Surgeon, specialty in oncology, Hospital General de México Dr. Eduardo Liceaga
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: DI/16/111/03/001
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Human Papillomavirus (HPV)-Related Cervical Cancer; HPV DNA
Keywords: CINtec Plus.; Pap test.; Progression to high-grade injury.; Xylo test.

STUDY DESIGN:
Intervention Model Description: Patients will be randomly selected by two sequences which will be used for diagnostic and positive patients will be referred for colposcopy and biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-test for cervical sample (Active Comparator): First sequence will start with self-test. Second sequence will start with traditional method.
  Interventions: Diagnostic Test: Cervical samples for identification of HR-HPV DNA via real-time PCTR.
- Traditional provider for cervical sample (Active Comparator): First sequence will start with traditional method. Second sequence will start with self-test method.
  Interventions: Diagnostic Test: Cervical samples for identification of HR-HPV DNA via real-time PCTR.

INTERVENTIONS:
Diagnostic Test: Cervical samples for identification of HR-HPV DNA via real-time PCTR. — Identification of HR-HPV DNA via real-time PCTR.

SUMMARY:
Problem Description When cervical cancer screening is needed, the Pap test (or Pap smears) is still the most common, although there are challenges that continue to prevent effective screening services in many countries, poor quality testing, long delays until screening is available, they give the results to women, poor population coverage and insufficient follow-up treatment. HPV testing can remove barriers related to access to screening services, since the woman can obtain the sample herself. Women's self-sampling for HPV testing has been used in a programmatic context in some countries. For a good impact, screening coverage must reach at least 70% of the target population. In the Region of the Americas, only seven countries have reported this level of coverage, so there is a great need for improvement.

Several factors make it difficult to improve coverage: most screening programs are unorganized, available mainly in urban areas, and based on the Pap test, which has been shown to have low sensitivity, limited and requires multiple consultations.

However, screening alone is not enough to prevent cervical cancer. Follow-up treatment of women with abnormal screening test results is necessary and remains a challenge.

Main objective To evaluate the effectiveness of cervicovaginal self-test in comparison with direct sampling by the service provider, for the identification of HR-HPV DNA via real-time PCTR and triage with dual staining biomarker p16 & ki67.

Methodology Under inclusion and exclusion criteria and signed informed consent, cervical sample will be taken with the corresponding method according to the randomization (self-test or service provider) and certify that the device did not cause damage or lacerations in the vaginal canal. In addition, an acceptability survey will be completed. All women with positive p16 & ki67 will be referred for colposcopy and biopsy. Patients will be informed her results with a specialist physician for guidance and indications.

Clinical study design is crossover, monocentric, randomized, open, and non-inferiority.

Statistical differences between self-test and service rpovider will be assesed.

DETAILED DESCRIPTION:
STUDY POPULATION The target population is patients admitted to HGM Oncology Service for cervical cancer screening through self-sampling and sampling by a service provider. Sample size is 444 valid patients

PROCESS Visit 1 is an inclusion visit. Participant will be included in the research protocol in accordance with the inclusion and exclusion criteria established by the protocol, and the signed informed consent will be collected. Patient will be randomized and sample will also be taken with the corresponding method and the patient will be completed to certify that the device did not cause damage or lacerations in the vaginal canal.

Visit 2 will be on the third day after taking the first sample. In this visit, the sample will be taken with the corresponding method according to the randomization and the patient will be completed to certify that the device did not cause damage or lacerations in the vaginal canal. In addition, the acceptability survey will be completed.

Visit 3 will take place 21 calendar days after the second visit, the results will be delivered to the patient, all women with positive results of CINtec Plus (p16 & ki67) will be referred for colposcopy and biopsy; said biopsies will be submitted for the analysis of over-expression of p16 protein. At this last visit, the patient will be informed of the importance and need to discuss her results with a specialist doctor for guidance and indications.

STATISTIC ANALYSIS The information to be analyzed are the results and the final diagnosis obtained by the self-test method (XytoTest device) and the service provider of the Oncology Service of the Hospital General de México "Eduardo Liceaga".

To determine the non-inferiority of both samples, the Kappa index will be used and to determine the significance through the Wilcoxon T.

ETHICAL AND BIOSAFETY ASPECTS The study complies with the ethical considerations corresponding to the 1964 Helsinki World Assembly and with their respective modifications in the World Medical Assembly, Hong Kong, September 1989 and Edinburgh, Scotland, October 2000 and the Clarification note of Paragraph 29, added by the General Assembly of the WMA, Washington 2002.

The informed consent format is authorized by the ethics and research committee and strictly adhere to the general health law and its regulations on research and the guidelines of the international conference on Harmonization (ICH) on good clinical practice ( GCP).

The subject is considered enrolled in the study when they have signed the informed consent form, no form must be completed or any research or study procedure must be completed before obtaining the written informed consent.

Any decision that might influence the subject's decision to remain in the study should be made known to investigator immediately.

Confidentiality of the subject will be maintained, all persons involved in the research who have access to the information, are obliged to refrain from disclosing the subject's information or any personal information.

This study is subject to be audited by Mexican regulatory authorities, with or without prior notice to the research site.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent
* Women with an active sex life
* Women 25 to 64 years old
* Patients without hysterectomy, conization of the cervix.
* Patients without radiotherapy treatment, cervical chemotherapy.
* 24 hours before taking the sample, they should not use douches, ovules, lubricants or gels.

Exclusion Criteria:

* Patients who have not started a sexual life
* Patients with uterine surgery.
* Patients pregnant.
* Patients with vaginal bleeding.
* Patients who have had sexual activity 24 hours prior to taking the sample.

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Cervical samples
Enrollment: 444 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
To assess effectiveness of cervicovaginal diagnosis by self-test in comparison with direct sampling by the service provider. | 5 months
  Identification of HPV-HR DNA via real-time PCTR and triage with dual-staining biomarker p16 & ki67.

SECONDARY OUTCOMES:
Acceptability for self-test | 5 months
  A survey will be applied to assess self-test acceptability in comparison to direct sampling by service provider

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Molina Fernández de Lara, PhD, Study Chair — Hospital General de México Eduardo Liceaga
Locations (1):
- Hospital General de México Eduardo Liceaga, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No